CLINICAL TRIAL: NCT00278408
Title: Randomized Study Comparing an Immuno-Chemotherapy With 6 Cycles of the Monoclonal Anti-CD20 Antibody Rituximab in Combination With 6 Cycles of Chemotherapy With CHOP ( Cyclophosphamide, Doxorubicin, Vincristine, and Prednisone) at 21-day Intervals or 14-day Intervals, Both With or Without Consolidating Radiotherapy or Large Tumour Masses (≥7.5 cm) and/or Extranodal Involvement in Patients With Aggressive CD20 B-Cell Lymphoma Aged 18 to 60 Years With Age-Adjusted IPI=1 (All) or IPI=0 With a Large Tumour Mass (≥7.5 cm) [UNFOLDER 21/14 Study]
Brief Title: Rituximab and Combination Chemotherapy With or Without Radiation Therapy in Treating Patients With B-Cell Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: German High-Grade Non-Hodgkin's Lymphoma Study Group (Other)
Responsible Party: Sponsor
Organization: Universität des Saarlandes (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000459796; DSHNHL-2004-3; EUDRACT-2005-005218-19; EU-205111
Record Dates: First submitted 2006-01-16; First posted 2006-01-18 (Estimated); Results first posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-05

CONDITIONS: Lymphoma
Keywords: contiguous stage II grade 3 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; stage I grade 3 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 3 follicular lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; stage I adult diffuse large cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; nodal marginal zone B-cell lymphoma; anaplastic large cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; contiguous stage II adult Burkitt lymphoma; contiguous stage II mantle cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II mantle cell lymphoma; stage I adult Burkitt lymphoma; stage I mantle cell lymphoma; stage III adult Burkitt lymphoma; stage III mantle cell lymphoma; stage IV adult Burkitt lymphoma; stage IV mantle cell lymphoma; contiguous stage II marginal zone lymphoma; noncontiguous stage II marginal zone lymphoma; stage I marginal zone lymphoma; stage III marginal zone lymphoma; stage IV marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Large-Cell, Anaplastic; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Lymphoma, Mantle-Cell | interventions — Filgrastim; Rituximab; Cyclophosphamide; Doxorubicin; Prednisone; Vincristine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Interventional: 6 R-CHOP-21 (Active Comparator): Arm I (R-CHOP-21): Patients receive R-CHOP immunochemotherapy comprising rituximab IV, cyclophosphamide IV over 15 minutes, doxorubicin IV, and vincristine IV on day 1 and oral prednisone once daily on days 1-5. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: rituximab; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: prednisone; Drug: vincristine sulfate
- Interventional: 6 R-CHOP-21 + radiotherapy (Active Comparator): Arm II (R-CHOP-21 and radiotherapy): Patients receive R-CHOP as in arm I. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Beginning 2-6 weeks after the last course of R-CHOP, patients who achieve a complete remission (CR) undergo radiotherapy 5 days a week for approximately 5½ weeks.
  Interventions: Biological: rituximab; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: prednisone; Drug: vincristine sulfate; Radiation: radiation therapy
- Interventional: 6 R-CHOP-14 (Active Comparator): Arm III (R-CHOP-14): Patients receive R-CHOP as in arm I. Patients also receive filgrastim (G-CSF) subcutaneously once daily on days 4-13 or until blood counts recover. Treatment repeats every 14 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: filgrastim; Biological: rituximab; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: prednisone; Drug: vincristine sulfate
- Interventional: 6 R-CHOP-14 and radiotherapy (Active Comparator): Arm IV (R-CHOP-14 and radiotherapy): Patients receive R-CHOP as in arm I. Patients also receive G-CSF an in arm III. Treatment repeats every 14 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Beginning 2-6 weeks after the last course of R-CHOP, patients who achieve CR undergo radiotherapy as in arm II.
  Interventions: Biological: filgrastim; Biological: rituximab; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: prednisone; Drug: vincristine sulfate; Radiation: radiation therapy

INTERVENTIONS:
Biological: filgrastim
  Arms: Interventional: 6 R-CHOP-14; Interventional: 6 R-CHOP-14 and radiotherapy
Biological: rituximab
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: prednisone
Drug: vincristine sulfate
Radiation: radiation therapy
  Arms: Interventional: 6 R-CHOP-14 and radiotherapy; Interventional: 6 R-CHOP-21 + radiotherapy

SUMMARY:
RATIONALE: Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some find cancer cells and kill them or carry cancer-killing substances to them. Others interfere with the ability of cancer cells to grow and spread. Drugs used in chemotherapy, such as cyclophosphamide, doxorubicin hydrochloride, vincristine, and prednisone, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill cancer cells. Giving rituximab and combination chemotherapy together with radiation therapy may kill more cancer cells. It is not yet known which schedule of rituximab and combination chemotherapy is more effective when given with or without radiation therapy in treating non-Hodgkin's lymphoma.

PURPOSE: This randomized phase III trial is studying two different schedules of rituximab and combination chemotherapy with or without radiation therapy to compare how well they work in treating patients with aggressive B-cell non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the time to treatment failure in patients with previously untreated, low-risk, aggressive, B-cell non-Hodgkin's lymphoma treated with 2 different schedules of immunochemotherapy comprising rituximab, cyclophosphamide, doxorubicin hydrochloride, vincristine, and prednisone with vs without radiotherapy.

Secondary

* Compare the time to progression in patients treated with these regimens.
* Compare the overall and disease-free/relapse-free survival of patients treated with these regimens.
* Compare the complete response rate in patients treated with these regimens.
* Compare the tumor control in patients treated with these regimens.
* Compare the safety of these regimens in these patients.
* Compare the pharmacoeconomics of these regimens.
* Compare patient adherence to these regimens.

OUTLINE: This is an open-label, randomized, multicenter study. Patients are stratified according to study center, serum lactic dehydrogenase level (≤ upper limit of normal [ULN] vs > ULN), disease stage (I or II vs III or IV), ECOG performance status (0-1 vs 2-3), bulky disease, and extranodal involvement. Patients with initial bulky disease and/or qualifying extranodal involvement are randomized to 1 of 4 treatment arms. Patients with non-bulky disease are randomized to treatment arms I or III.

All patients will be given the option of receiving a 1-week course of pretreatment therapy comprising vincristine IV once on day -6 and oral prednisone once daily on days -6 to 0.

* Arm I (R-CHOP-21): Patients receive R-CHOP immunochemotherapy comprising rituximab IV, cyclophosphamide IV over 15 minutes, doxorubicin IV, and vincristine IV on day 1 and oral prednisone once daily on days 1-5. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
* Arm II (R-CHOP-21 and radiotherapy): Patients receive R-CHOP as in arm I. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Beginning 2-6 weeks after the last course of R-CHOP, patients who achieve a complete remission (CR) undergo radiotherapy 5 days a week for approximately 5½ weeks.
* Arm III (R-CHOP-14): Patients receive R-CHOP as in arm I. Patients also receive filgrastim (G-CSF) subcutaneously once daily on days 4-13 or until blood counts recover. Treatment repeats every 14 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
* Arm IV (R-CHOP-14 and radiotherapy): Patients receive R-CHOP as in arm I. Patients also receive G-CSF an in arm III. Treatment repeats every 14 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Beginning 2-6 weeks after the last course of R-CHOP, patients who achieve CR undergo radiotherapy as in arm II.

Patients in all arms undergo restaging of their disease after courses 3 and 6 of R-CHOP. Patients with stable disease after 6 courses or disease progression after courses 3 or 6 proceed to salvage chemotherapy off study. Patients achieving a partial remission or an unconfirmed CR after 6 courses undergo additional restaging 4 weeks later. Patients with disease progression proceed to salvage chemotherapy off study. Patients who achieve CR after 6 courses of R-CHOP or have a confirmed CR after the additional restaging undergo radiotherapy according to randomization (as above).

After completion of study treatment, patients are followed periodically for 5 years and then annually thereafter.

PROJECTED ACCRUAL: A total of 1,072 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed aggressive B-cell non-Hodgkin's lymphoma, including the following subtypes:

  * Grade 3 follicular lymphoma
  * Diffuse B-cell lymphoma, including diffuse large cell lymphoma with the following variants:

    * Centroblastic
    * Immunoblastic
    * Plasmablastic
    * Anaplastic large cell
    * T-cell-rich B-cell lymphoma
  * Primary effusion lymphoma
  * Intravascular B-cell lymphoma
  * Primary mediastinal B-cell lymphoma
  * Burkitt's or Burkitt-like lymphoma
  * Mantle cell lymphoma (blastoid)
  * Aggressive marginal zone lymphoma (monocytoid)
* Previously untreated disease
* CD20-positive disease
* International prognostic index (IPI) score 0 or 1 (age-adjusted)

  * Only patients with bulky disease, as defined by largest single or conglomerate tumor ≥ 7.5 cm in diameter, are allowed to have an IPI score of 0
* No mucosa-associated lymphoid tissue (MALT) lymphoma
* No CNS involvement of lymphoma (intracerebral, meningeal, or intraspinal)

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Platelet count ≥ 100,000/mm³
* WBC ≥ 2,500/mm³
* No known hypersensitivity to the study medications
* No known HIV-positivity
* No active hepatitis infection
* Not pregnant or lactating
* Negative pregnancy test
* No other malignancy within the past 5 years except carcinoma in situ or basal cell skin cancer
* No impaired left ventricular function
* No severe cardiac arrhythmias
* No other impaired organ function
* No other serious disorder

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy or radiotherapy
* No prior immunosuppressive treatment with cytostatics
* No concurrent participation in other treatment studies

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 700 (Actual)
Dates: Start 2006-01-02; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael G.M. Pfreundschuh, MD †, Study Chair — Universitaetsklinikum des Saarlandes; Viola Poeschel, MD, Study Director — Study Office Homburg
Locations (152):
- Denmark (2):
  - Rigshospitalet, Department of Hematology, Copenhagen
  - Amtssygehuset i Herlev, Herlev
- Germany (138):
  - GMP Tummes/Weinberg, Aachen
  - Klinikum St. Marien, Amberg
  - Klinikum Augsburg, Augsburg
  - Kreiskrankenhaus Aurich, Aurich
  - Klinikum Bayreuth, Bayreuth
  - Charite - Campus Charite Mitte, Berlin
  - Charite University Hospital - Campus Virchow Klinikum, Berlin
  - Helios Klinikum Berlin-Buch, Department of Hematology and Stem Cell Transplantation, Berlin
  - Franziskus Hospital, Bielefeld
  - Augusta-Kranken-Anstalt gGmbH, Bochum
  - Johanniter Krankenhaus Bonn, Bonn
  - Universitätsklinikum Bonn, Bonn
  - Staedtisches Klinikum Braunschweig, Braunschweig
  - Klinikum Bremen-Mitte, Bremen
  - Evangelisches Diakonie-Krankenhaus gGmbH, Department of Internal Medicine, Bremen
  - Praxis Dr. Obst, Burgwedel
  - Onkologische Schwerpunktpraxis Celle, Celle
  - Hospital Kuchwald Chemnitz - Department of Internal Medicine III, Chemnitz
  - Klinikum Chemnitz, Chemnitz
  - Klinikum Coburg, Coburg
  - Praxis Fuer Haematologie Internistische Onkologie, Cologne
  - Medizinische Universitaetsklinik I at the University of Cologne, Cologne
  - Gemeinschaftspraxis Dres. Schmitz, Steinmetz, Severin, Cologne
  - Krankenhaus Holweide, Cologne
  - Lungenklinik Köln-Merheim, Cologne
  - Carl - Thiem - Klinkum Cottbus, Cottbus
  - Klinikum Dortmund, Dortmund
  - Virngrund-Klinik Ellwangen, Ellwangen
  - Hans - Susemihl - Krankenhaus, Emden
  - Universitätsklinikum Erlangen, Erlangen
  - St. Antonius Hospital, Eschweiler
  - Universitaetsklinikum Essen, Essen
  - Klinikum Esslingen, Esslingen am Neckar
  - Krankenhaus Nordwest, Frankfurt
  - Klinikum der J.W. Goethe Universitaet, Frankfurt
  - Klinikum Frankfurt (Oder) GmbH, Frankfurt (Oder)
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - GMP Dres. Marschner, Zaiss, Kirste, Semsek, Freiburg im Breisgau
  - Praxis Dr. med. Reiber, Freiburg im Breisgau
  - Klinikum Fulda, Fulda
  - Klinikum Garmisch - Partenkirchen GmbH, Garmisch-Partenkirchen
  - Saint Josef Hospital, Gelsenkirchen
  - Praxis Dr. med. Schliesser, Giessen
  - Wilhelm-Anton-Hospital gGmbH, Goch, Goch
  - Universitaetsklinikum Goettingen, Department of Hematology and Oncology, Göttingen
  - Klinik Fuer Innere Medizin, Hematology/Oncology, Ernst Moritz Armdt Universitaet, Greifswald
  - Gemeinschaftspraxis, Güstrow
  - St. Marien Hospital - Katholisches Krankenhaus Hagen gGmbH, Hagen
  - Krankenhaus Martha-Maria Halle-Doelau gGmbH, Halle
  - GMP Rohrberg, Hurtz, Schmidt, Frank-Gleich, Halle
  - Asklepios Klinik St. Georg, Hamburg
  - University Medical Center Hamburg - Eppendorf, Hamburg
  - Hämatologisch-onkologische Praxis Altona (HOPA), Hamburg
  - Evangelisches Krankenhaus Hamm, Hamm
  - Klinikum Stadt Hanau, Hanau
  - Krankenhaus Siloah - Medizinische Klinik II, Hanover
  - Medizinische Hochschule Hannover, Hanover
  - Medizinische Universitaetsklinik und Poliklinik, Heidelberg
  - Klinikum Kreis Herford, Herford
  - Privatklinik Dr. R. Schindlbeck GmbH & Co. KG, Herrsching am Ammersee
  - St. Bernward Krankenhaus, Hildesheim
  - Evangelisches Krankenhaus Holzminden, Holzminden
  - Haematologie und Internistische Onkologie Praxis, Homberg (Efze)
  - Universitaetsklinikum des Saarlandes, Homburg
  - Clinic for Bone Marrow Transplantation and Hematology and Oncology, Idar-Oberstein
  - Staedtisches Klinikum Karlsruhe gGmbH, Karlsruhe
  - St. Vincentius Kliniken Karlsruhe, Karlsruhe
  - Internistische Gemeinschaftspraxis - Kassel, Kassel
  - Klinikum Kempten Oberallgaeu, Kempten
  - Staedtisches Krankenhaus Kiel, Kiel
  - University Hospital Schleswig-Holstein - Kiel Campus, Kiel
  - Gemeinschaftspraxis Dres. Heymanns, Weide, Thomalla, Koblenz
  - Praxis Dr. Stauch, Kronach
  - Internistische Praxis - Landshut, Landshut
  - Klinikum Landshut, Landshut
  - Caritas Krankenhaus Lebach, Lebach
  - Onkologische Schwerpunktpraxis Dr. Lothar Müller, Leer
  - Klinikum St. Georg Leipzig, Leipzig
  - Onkologische Praxis am Diakonissenhaus, Leipzig
  - Klinikum Lippe-Lemgo, Lemgo
  - St. Marienkrankenhaus, Ludwigshafen
  - Klinikum der Stadt Ludwigshafen am Rhein, Ludwigshafen am Rhein
  - Universitätsklinikum Schleswig-Holstein, Lübeck
  - Kreiskrankenhaus Luedenscheid, Lüdenscheid
  - Universitaetsklinkum Magdeburg der Otto-von-Guericke-Universitaet Magdeburg, Magdeburg
  - Krankenhaus Altstadt Magdeburg, Magdeburg
  - III Medizinische Klinik Mannheim, Mannheim
  - Mannheimer Onkologie Praxis, Mannheim
  - Universitätsklinikum Gießen und Marburg (UKGM), Marburg
  - Klinikum Minden, Minden
  - Krankenhaus Maria Hilf GmbH, Mönchengladbach
  - Klinikum der Universitaet Muenchen - Grosshadern Campus, Munich
  - Klinikum Rechts Der Isar - Technische Universitaet Muenchen, Munich
  - Gemeinschaftspraxis Abenhardt, Bojko, Bosse, Riedner, Munich
  - Städtisches Klinikum München Harlaching, Munich
  - Stauferklinikum Schwäbisch Gmünd, Mutlangen
  - Gemeinschaftspraxis Dres. Schröder, Sieg, Mülheim
  - Haematologisch - Onkologische Gemeinschaftspraxis - Muenster, Münster
  - Medizinische Klinik und Poliklinik A - Universitaetsklinikum Muenster, Münster
  - Onkologische Schwerwpunktpraxis Dr. Ladda, Neumarkt
  - Lukaskrankenhaus Neuss, Neuss
  - BRK Schloßbergklinik Oberstaufen, Oberstaufen
  - GMP Dres. Balló, Böck, Offenbach
  - Klinikum Oldenburg - Department of Hematology and Oncology, Oldenburg
  - Pius Hospital Oldenburg, Department of Internal Oncology, Oldenburg
  - Paracelsus Krankenhaus Ruit, Ostfildern
  - Bruederkrankenhaus St. Josef Paderborn, Paderborn
  - Krankenhaus Siloah, Pforzheim
  - Praxis Dr. Dencausse, Pforzheim
  - Klinikum der Universitaet Regensburg, Regensburg
  - Krankenhaus Barmherzige Brüder Regensburg, Regensburg
  - Klinikum am Steinenberg, Reutlingen
  - Klinikum Suedstadt Rostock, Rostock
  - Universitätsklinikum Rostock, Rostock
  - Gemeinschaftspraxis Dres. Jacobs, Daus, Schmits, Saarbrücken
  - Leopoldina - Krankenhaus, Schweinfurt
  - St. Marien - Krankenhaus Siegen GMBH, Siegen
  - Onkologische Schwerpunktpraxis - Straubing, Straubing
  - Klinik fuer Onkologie - Katharinenhospital Stuttgart, Stuttgart
  - Diakonie Klinikum Stuttgart, Stuttgart
  - Bürgerhospital, Stuttgart
  - Krankenanstalt Mutterhaus der Borromaerinnen, Trier
  - Krankenhaus Der Barmherzigen Brueder, Trier
  - Praxis Fuer Internistische Haematologie / Onkologie, Troisdorf
  - Universitätsklinikum Tübingen, Department of Internal Medicine II, Tübingen
  - Praxis fuer Haematologie und Onkologie, Twistringen
  - Comprehensive Cancer Center Ulm at Universitaetsklinikum Ulm, Ulm
  - Katharinen Hospital Unna, Unna
  - St. Marienhospital - Vechta, Vechta
  - Praxis VS-Villingen, Villingen-Schwenningen
  - Regional Hospital Waldbrol, Waldbröl
  - Med. Versorgungszentrum Weiden, Weiden
  - Harz-Klinikum-Wernigerode, Wernigerode
  - Ammerland Klinik GmbH Westerstede, Westerstede
  - Dr. Horst-Schmidt-Kliniken, Wiesbaden
  - Kliniken St. Antonius, Wuppertal
  - Helios Klinikum Wuppertal, Wuppertal
  - Heinrich-Braun-Krankenhaus Zwickau, Zwickau
- Rabin Medical Center - Beilinson Campus, Petah Tikva, Israel
- Italy (11):
  - Ospidale A. Cardarelli, Campobasso
  - Azienda Ospedaliera di Cosenza, Cosenza
  - AOU San Martino Genova, Genova
  - Az. Ospedaliera Messina, Messina
  - Policlinico Universitario "G. Martino" Messina, Messina
  - Centro Oncologico Modenese, University of Modena and Reggio Emilia, Modena
  - Ematologia - OSP. Civile Piacenza, Piacenza
  - A. Santa Maria Nuova, Hematology Azienda, Reggio Emilia
  - Osp. S. Vincenzo - Taormina, Taormina
  - Ospedale San Giuseppe Moscati, Taranto
  - Ospedale di circolo e Fondazione Macchi Varese, Varese

REFERENCES:
- [Result] Radiotherapy (RT) to bulky (B) and extralymphatic (E) disease in combination with 6xR-CHOP-14 or R-CHOP-21 in young good-prognosis DLBCL patients: Results of the 2x2 randomized UNFOLDER trial of the DSHNHL/GLA. Michael Pfreundschuh, Niels Murawski, Marita Ziepert, Bettina Altmann, Martin H. Dreyling, Peter Borchmann, Stefano Luminari, Mathias Witzens-Harig, Judith Dierlamm, Mathias Haenel, Lorenz Truemper, Bernd Metzner, Eva Lengfelder, Ulrich B. Keller, Christian Ruebe, Christian Berdel, Norbert Schmitz, Gerhard Held, and Viola Poeschel Journal of Clinical Oncology 2018 36:15_suppl, 7574-7574
- [Result] Role of radiotherapy and dose-densification of R-CHOP in primary mediastinal B-cell lymphoma: A subgroup analysis of the unfolder trial of the German Lymphoma Alliance (GLA). Gerhard Held, Lorenz Thurner, Viola Poeschel, Christian Berdel, German Ott, Christian Schmidt, Andreas Viardot, Peter Borchmann, Ofer Shpilberg, Maike Nickelsen, Massimo Federico, Peter de Nully Brown, Niels Murawski, Lorenz H. Trumper, Heinz Schmidberger, Christian Ruebe, Jochen Fleckenstein, Norbert Schmitz, Markus Loeffler, Marita Ziepert, and German Lymphoma Alliance Journal of Clinical Oncology 2020 38:15_suppl, 8041-8041
- [Derived] Thurner L, Ziepert M, Berdel C, Schmidt C, Borchmann P, Kaddu-Mulindwa D, Viardot A, Witzens-Harig M, Dierlamm J, Haenel M, Metzner B, Wulf G, Lengfelder E, Keller UB, Frickhofen N, Nickelsen M, Gaska T, Griesinger F, Mahlberg R, Marks R, Shpilberg O, Lindemann HW, Soekler M, Fischer von Weikersthal L, Kiehl M, Roemer E, Bentz M, Krammer-Steiner B, Trappe R, de Nully Brown P, Federico M, Merli F, Engelhard M, Glass B, Schmitz N, Truemper L, Bewarder M, Hartmann F, Murawski N, Stilgenbauer S, Rosenwald A, Altmann B, Schmidberger H, Fleckenstein J, Loeffler M, Poeschel V, Held G. Radiation and Dose-densification of R-CHOP in Aggressive B-cell Lymphoma With Intermediate Prognosis: The UNFOLDER Study. Hemasphere. 2023 Jul 5;7(7):e904. doi: 10.1097/HS9.0000000000000904. eCollection 2023 Jul. PMID 37427146

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 02nd January 2006, to 16th November 2015, 700 patients were enrolled at 148 sites including hospitals and private practitioners.
Groups:
- Interventional: 6 R-CHOP-21 for Patients With Radiotherapy Indication: Arm I (R-CHOP-21): Patients receive R-CHOP immunochemotherapy comprising rituximab IV, cyclophosphamide IV over 15 minutes, doxorubicin IV, and vincristine IV on day 1 and oral prednisone once daily on days 1-5. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  rituximab
  cyclophosphamide
  doxorubicin hydrochloride
  prednisone
  vincristine sulfate
- Interventional: 6 R-CHOP-14 for Patients With Radiotherapy Indication: Arm II (R-CHOP-14): Patients receive R-CHOP immunochemotherapy comprising rituximab IV, cyclophosphamide IV over 15 minutes, doxorubicin IV, and vincristine IV on day 1 and oral prednisone once daily on days 1-5. Treatment repeats every 14 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  rituximab
  cyclophosphamide
  doxorubicin hydrochloride
  prednisone
  vincristine sulfate
  filgrastim
- Interventional: 6 R-CHOP-21 + Radiotherapy for Patients With Radiotherapy Indication: Arm III (R-CHOP-21): Patients receive R-CHOP immunochemotherapy comprising rituximab IV, cyclophosphamide IV over 15 minutes, doxorubicin IV, and vincristine IV on day 1 and oral prednisone once daily on days 1-5. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity followed by consolidating radiotherapy with 39.6 Gy.
  rituximab
  cyclophosphamide
  doxorubicin hydrochloride
  prednisone
  vincristine sulfate
- Interventional: 6 R-CHOP-14 + Radiotherapy for Patients With Radiotherapy Indication: Arm IV (R-CHOP-14): Patients receive R-CHOP immunochemotherapy comprising rituximab IV, cyclophosphamide IV over 15 minutes, doxorubicin IV, and vincristine IV on day 1 and oral prednisone once daily on days 1-5. Treatment repeats every 14 days for up to 6 courses in the absence of disease progression or unacceptable toxicity followed by consolidating radiotherapy with 39.6 Gy.
  rituximab
  cyclophosphamide
  doxorubicin hydrochloride
  prednisone
  vincristine sulfate
  filgrastim
- Interventional: 6 R-CHOP-21 for Patients Without Radiotherapy Indication: Arm V (R-CHOP-21): Patients receive R-CHOP immunochemotherapy comprising rituximab IV, cyclophosphamide IV over 15 minutes, doxorubicin IV, and vincristine IV on day 1 and oral prednisone once daily on days 1-5. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  rituximab
  cyclophosphamide
  doxorubicin hydrochloride
  prednisone
  vincristine sulfate
- Interventional: 6 R-CHOP-14 for Patients Without Radiotherapy Indication: Arm VI (R-CHOP-14): Patients receive R-CHOP immunochemotherapy comprising rituximab IV, cyclophosphamide IV over 15 minutes, doxorubicin IV, and vincristine IV on day 1 and oral prednisone once daily on days 1-5. Treatment repeats every 14 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  rituximab
  cyclophosphamide
  doxorubicin hydrochloride
  prednisone
  vincristine sulfate
  filgrastim
Period: Overall Study
Arm/Group | Interventional: 6 R-CHOP-21 for Patients With Radiotherapy Indication | Interventional: 6 R-CHOP-14 for Patients With Radiotherapy Indication | Interventional: 6 R-CHOP-21 + Radiotherapy for Patients With Radiotherapy Indication | Interventional: 6 R-CHOP-14 + Radiotherapy for Patients With Radiotherapy Indication | Interventional: 6 R-CHOP-21 for Patients Without Radiotherapy Indication | Interventional: 6 R-CHOP-14 for Patients Without Radiotherapy Indication
Started | 81 | 81 | 155 | 150 | 114 | 114
Completed | 77 | 79 | 133 | 135 | 110 | 109
Not Completed | 4 | 2 | 22 | 15 | 4 | 5

BASELINE CHARACTERISTICS:
Population: 700 patients were randomized, however 695 were analyzed due to a withdrawal of consent (5 patients)
Groups:
- Total: Total of all reporting groups
Arm/Group | Interventional: 6 R-CHOP-21 for Patients With Radiotherapy Indication | Interventional: 6 R-CHOP-14 for Patients With Radiotherapy Indication | Interventional: 6 R-CHOP-21 + Radiotherapy for Patients With Radiotherapy Indication | Interventional: 6 R-CHOP-14 + Radiotherapy for Patients With Radiotherapy Indication | Interventional: 6 R-CHOP-21 for Patients Without Radiotherapy Indication | Interventional: 6 R-CHOP-14 for Patients Without Radiotherapy Indication | Total
Number analyzed (Participants) | 81 | 81 | 155 | 150 | 114 | 114 | 695
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 81 | 81 | 155 | 150 | 114 | 114 | 695
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 43 [20 to 60] | 45 [20 to 60] | 46 [18 to 60] | 44 [18 to 60] | 50 [18 to 60] | 49 [20 to 60] | 47 [18 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 38 | 69 | 67 | 43 | 43 | 292
  Male | 49 | 43 | 86 | 83 | 71 | 71 | 403
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: 3 Years Event-free Survival
Description: Event-free survival was the primary endpoint, which was defined as the time from randomization until one of the following events had occurred: progression during therapy, partial response, no change, unknown status at the end of study therapy, relapse after complete response or unconfirmed complete response, death from any cause; or additional treatment, whichever came first.
Time Frame: Each patient will be observed for 3 years starting from completion of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Interventional: 6 R-CHOP-21 for Patients With Radiotherapy Indication | Interventional: 6 R-CHOP-14 for Patients With Radiotherapy Indication | Interventional: 6 R-CHOP-21 + Radiotherapy for Patients With Radiotherapy Indication | Interventional: 6 R-CHOP-14 + Radiotherapy for Patients With Radiotherapy Indication | Interventional: 6 R-CHOP-21 for Patients Without Radiotherapy Indication | Interventional: 6 R-CHOP-14 for Patients Without Radiotherapy Indication
Number analyzed (Participants) | 81 | 81 | 155 | 150 | 114 | 114
Participants | 51 | 56 | 126 | 123 | 89 | 92

2. Secondary Outcome: 3 Years Progression-free Survival
Description: Progression of disease is defined as: recurrence of disease symptoms, development of new lymphatic or extralymphatic lesions or marked increase in lymphoma manifestation size by more than 25% in comparison with baseline.
Time Frame: Each patient will be observed for 3 years starting from completion of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Interventional: 6 R-CHOP-21 for Patients With Radiotherapy Indication | Interventional: 6 R-CHOP-14 for Patients With Radiotherapy Indication | Interventional: 6 R-CHOP-21 + Radiotherapy for Patients With Radiotherapy Indication | Interventional: 6 R-CHOP-14 + Radiotherapy for Patients With Radiotherapy Indication | Interventional: 6 R-CHOP-21 for Patients Without Radiotherapy Indication | Interventional: 6 R-CHOP-14 for Patients Without Radiotherapy Indication
Number analyzed (Participants) | 81 | 81 | 155 | 150 | 114 | 114
Participants | 64 | 68 | 133 | 136 | 96 | 104

3. Secondary Outcome: 3 Years Overall Survival
Description: Overall survival was defined as the time from randomization to death of any cause.
Time Frame: Each patient will be observed for 3 years starting from completion of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Interventional: 6 R-CHOP-21 for Patients With Radiotherapy Indication | Interventional: 6 R-CHOP-14 for Patients With Radiotherapy Indication | Interventional: 6 R-CHOP-21 + Radiotherapy for Patients With Radiotherapy Indication | Interventional: 6 R-CHOP-14 + Radiotherapy for Patients With Radiotherapy Indication | Interventional: 6 R-CHOP-21 for Patients Without Radiotherapy Indication | Interventional: 6 R-CHOP-14 for Patients Without Radiotherapy Indication
Number analyzed (Participants) | 81 | 81 | 155 | 150 | 114 | 114
Participants | 76 | 74 | 144 | 141 | 107 | 108

4. Secondary Outcome: Rate of Complete Remissions and Progressive Disease
Time Frame: Each patient will be observed for 3 years starting from completion of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Interventional: 6 R-CHOP-21 for Patients With Radiotherapy Indication | Interventional: 6 R-CHOP-14 for Patients With Radiotherapy Indication | Interventional: 6 R-CHOP-21 + Radiotherapy for Patients With Radiotherapy Indication | Interventional: 6 R-CHOP-14 + Radiotherapy for Patients With Radiotherapy Indication | Interventional: 6 R-CHOP-21 for Patients Without Radiotherapy Indication | Interventional: 6 R-CHOP-14 for Patients Without Radiotherapy Indication
Number analyzed (Participants) | 81 | 81 | 155 | 150 | 114 | 114
Participants
  Rate of complete remissions | 64 | 64 | 141 | 133 | 109 | 105
  Rate of progressive disease | 4 | 2 | 4 | 6 | 1 | 0

5. Secondary Outcome: Number of Patients With a Relapse After a CR/CRu
Description: Relapse is defined as, recurrence of disease symptoms, development of new lymphatic or extralymphatic lesions or a marked increase in lymphoma manifestation size by more thyn 25% after at least 2 months CR or CRu from the time point of the final restaging examination
Time Frame: Each patient will be observed for 3 years starting from completion of treatment.
Population: Only patients who reached a CR/CRu after at least 2 months after the final restaging examination were taken for the relapse analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Interventional: 6 R-CHOP-21 for Patients With Radiotherapy Indication | Interventional: 6 R-CHOP-14 for Patients With Radiotherapy Indication | Interventional: 6 R-CHOP-21 + Radiotherapy for Patients With Radiotherapy Indication | Interventional: 6 R-CHOP-14 + Radiotherapy for Patients With Radiotherapy Indication | Interventional: 6 R-CHOP-21 for Patients Without Radiotherapy Indication | Interventional: 6 R-CHOP-14 for Patients Without Radiotherapy Indication
Number analyzed (Participants) | 64 | 64 | 142 | 133 | 110 | 105
Participants | 12 | 8 | 13 | 9 | 18 | 7

6. Secondary Outcome: Safety (Adverse Events, Serious Adverse Events, Rate of Secondary Neoplasia, Selected Laboratory Parameters, Including Leucocytes, Thrombocytes, and Haemoglobin)
Time Frame: Each patient will be observed for 3 years starting from completion of treatment.
Population: The number analyzed differs from overall number analyzed due to missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | Interventional: 6 R-CHOP-21 for Patients With Radiotherapy Indication | Interventional: 6 R-CHOP-14 for Patients With Radiotherapy Indication | Interventional: 6 R-CHOP-21 + Radiotherapy for Patients With Radiotherapy Indication | Interventional: 6 R-CHOP-14 + Radiotherapy for Patients With Radiotherapy Indication | Interventional: 6 R-CHOP-21 for Patients Without Radiotherapy Indication | Interventional: 6 R-CHOP-14 for Patients Without Radiotherapy Indication
Number analyzed (Participants) | 81 | 81 | 155 | 150 | 114 | 114
Participants
  rate of secondary neoplasm | 4 | 1 | 7 | 4 | 8 | 8
  Leukocytopenia CTC 3 - 4: number analyzed (Participants) | 43 | 44 | 76 | 83 | 49 | 55
  Leukocytopenia CTC 3 - 4 | 31 | 22 | 45 | 36 | 21 | 21
  Thrombocytopenia CTC 3 - 4: number analyzed (Participants) | 76 | 75 | 142 | 137 | 99 | 103
  Thrombocytopenia CTC 3 - 4 | 3 | 3 | 3 | 0 | 2 | 1
  Anemia CTC 3 - 4: number analyzed (Participants) | 76 | 76 | 145 | 136 | 100 | 104
  Anemia CTC 3 - 4 | 1 | 3 | 9 | 10 | 2 | 11
  Nausea CTC 3 - 5: number analyzed (Participants) | 75 | 75 | 148 | 138 | 105 | 112
  Nausea CTC 3 - 5 | 1 | 5 | 7 | 5 | 1 | 3
  Vomiting CTC 3 - 5: number analyzed (Participants) | 74 | 75 | 148 | 137 | 105 | 112
  Vomiting CTC 3 - 5 | 1 | 3 | 4 | 2 | 2 | 1
  Diarrhoe CTC 3 - 5: number analyzed (Participants) | 76 | 75 | 149 | 139 | 105 | 112
  Diarrhoe CTC 3 - 5 | 0 | 1 | 2 | 1 | 0 | 1
  Constipation CTC 3 - 5: number analyzed (Participants) | 75 | 74 | 148 | 139 | 105 | 112
  Constipation CTC 3 - 5 | 1 | 0 | 2 | 2 | 0 | 2
  Mucositis CTC 3 - 5: number analyzed (Participants) | 76 | 75 | 149 | 140 | 105 | 112
  Mucositis CTC 3 - 5 | 0 | 1 | 0 | 1 | 0 | 3
  Arrhythmia CTC 3 - 5: number analyzed (Participants) | 75 | 74 | 149 | 141 | 105 | 112
  Arrhythmia CTC 3 - 5 | 0 | 0 | 0 | 2 | 2 | 0
  Cardiac functions CTC 3 - 5: number analyzed (Participants) | 73 | 72 | 149 | 138 | 105 | 112
  Cardiac functions CTC 3 - 5 | 0 | 0 | 1 | 2 | 0 | 0
  Sensory CTC 3 - 5: number analyzed (Participants) | 75 | 76 | 150 | 141 | 103 | 111
  Sensory CTC 3 - 5 | 3 | 4 | 10 | 4 | 3 | 8
  Mood CTC 3 - 5: number analyzed (Participants) | 74 | 75 | 148 | 139 | 105 | 112
  Mood CTC 3 - 5 | 0 | 0 | 1 | 0 | 0 | 1
  Allergy CTC 3 - 5: number analyzed (Participants) | 75 | 75 | 149 | 139 | 105 | 113
  Allergy CTC 3 - 5 | 2 | 4 | 1 | 3 | 0 | 1
  Infection CTC 3 - 5: number analyzed (Participants) | 79 | 78 | 152 | 144 | 105 | 113
  Infection CTC 3 - 5 | 6 | 12 | 13 | 15 | 8 | 12

7. Secondary Outcome: Adherence to Protocol - Absolute Dose Vincristine and Prednisone in mg (Median)
Time Frame: Each patient will be observed for 3 years starting from completion of treatment.
Measure: Median (Full Range); unit: mg
Arm/Group | Interventional: 6 R-CHOP-21 for Patients With Radiotherapy Indication | Interventional: 6 R-CHOP-14 for Patients With Radiotherapy Indication | Interventional: 6 R-CHOP-21 + Radiotherapy for Patients With Radiotherapy Indication | Interventional: 6 R-CHOP-14 + Radiotherapy for Patients With Radiotherapy Indication | Interventional: 6 R-CHOP-21 for Patients Without Radiotherapy Indication | Interventional: 6 R-CHOP-14 for Patients Without Radiotherapy Indication
Number analyzed (Participants) | 81 | 81 | 155 | 150 | 114 | 114
mg
  Absolute dose vincristine | 12 [2 to 13] | 12 [2 to 12] | 12 [2 to 13] | 12 [4 to 12] | 12 [2 to 12] | 12 [2 to 12]
  Absolute dose prednisone | 3000 [500 to 5750] | 3000 [400 to 3750] | 3000 [500 to 3900] | 3000 [1000 to 3900] | 3000 [1000 to 6000] | 3000 [500 to 4000]

8. Secondary Outcome: Health-economic Aspects - Number of Patients Who Received Antibiotic Intervention and/or Red Blood Cell and Platelet Transfusion
Time Frame: Each patient will be observed for 3 years starting from completion of treatment.
Population: The number analyzed differs from overall number analyzed due to missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | Interventional: 6 R-CHOP-21 for Patients With Radiotherapy Indication | Interventional: 6 R-CHOP-14 for Patients With Radiotherapy Indication | Interventional: 6 R-CHOP-21 + Radiotherapy for Patients With Radiotherapy Indication | Interventional: 6 R-CHOP-14 + Radiotherapy for Patients With Radiotherapy Indication | Interventional: 6 R-CHOP-21 for Patients Without Radiotherapy Indication | Interventional: 6 R-CHOP-14 for Patients Without Radiotherapy Indication
Number analyzed (Participants) | 81 | 81 | 155 | 150 | 114 | 114
Participants
  antibiotics interventional per patient: number analyzed (Participants) | 79 | 80 | 154 | 147 | 105 | 113
  antibiotics interventional per patient | 21 | 25 | 42 | 39 | 22 | 36
  red blood cell and platelet transfusions per patient: number analyzed (Participants) | 80 | 79 | 154 | 147 | 105 | 113
  red blood cell and platelet transfusions per patient | 1 | 9 | 5 | 14 | 4 | 16

9. Secondary Outcome: Adherence to Protocol - Total Duration of Chemotherapy in Days (Median)
Time Frame: Each patient will be observed for 3 years starting from completion of treatment.
Measure: Median (Full Range); unit: days
Arm/Group | Interventional: 6 R-CHOP-21 for Patients With Radiotherapy Indication | Interventional: 6 R-CHOP-14 for Patients With Radiotherapy Indication | Interventional: 6 R-CHOP-21 + Radiotherapy for Patients With Radiotherapy Indication | Interventional: 6 R-CHOP-14 + Radiotherapy for Patients With Radiotherapy Indication | Interventional: 6 R-CHOP-21 for Patients Without Radiotherapy Indication | Interventional: 6 R-CHOP-14 for Patients Without Radiotherapy Indication
Number analyzed (Participants) | 81 | 81 | 155 | 150 | 114 | 114
days | 105 [20 to 126] | 70 [69 to 99] | 105 [102 to 124] | 71 [14 to 111] | 105 [21 to 137] | 70 [14 to 112]

10. Secondary Outcome: Adherence to Protocol - Absolute Dose Cyclophosphamide, Doxorubicin and Rituximab in mg/m² (Median)
Time Frame: Each patient will be observed for 3 years starting from completion of treatment.
Measure: Median (Full Range); unit: mg/m²
Arm/Group | Interventional: 6 R-CHOP-21 for Patients With Radiotherapy Indication | Interventional: 6 R-CHOP-14 for Patients With Radiotherapy Indication | Interventional: 6 R-CHOP-21 + Radiotherapy for Patients With Radiotherapy Indication | Interventional: 6 R-CHOP-14 + Radiotherapy for Patients With Radiotherapy Indication | Interventional: 6 R-CHOP-21 for Patients Without Radiotherapy Indication | Interventional: 6 R-CHOP-14 for Patients Without Radiotherapy Indication
Number analyzed (Participants) | 81 | 81 | 155 | 150 | 114 | 114
mg/m²
  Cyclophosphamide | 4474 [750 to 4693] | 4482 [738 to 4875] | 4464 [762 to 4750] | 4474 [1480 to 4667] | 4476 [1364 to 4737] | 4455 [742 to 4714]
  Doxorubicin | 300 [50 to 316] | 300 [50 to 323] | 299 [48 to 316] | 298 [90 to 314] | 298 [91 to 318] | 298 [50 to 314]
  Rituximab | 2244 [350 to 2438] | 2232 [375 to 2413] | 2238 [371 to 2500] | 2245 [740 to 2402] | 2242 [682 to 2520] | 2228 [389 to 2471]

ADVERSE EVENTS:
Time Frame: Each patient will be observed for at least 3 years starting from completion of treatment.
Description: Please note that all patients (pts) had suffered from, at least, one non-SAE. We entered the no. of pts who could have suffered from non-SAEs of CTC-Gr. 3-5 (=no. of pts randomized in each arm), as this was the only part of the non-SAEs, which were statistically analysed. Multiple counts have been possible, as pts could have suffered from more than one non-SAE of CTC-Gr. 3-5.
  The number analyzed differs from overall number analyzed due to missing data.
Arm/Group | Interventional: 6 R-CHOP-21 for Patients With Radiotherapy Indication | Interventional: 6 R-CHOP-14 for Patients With Radiotherapy Indication | Interventional: 6 R-CHOP-21 + Radiotherapy for Patients With Radiotherapy Indication | Interventional: 6 R-CHOP-14 + Radiotherapy for Patients With Radiotherapy Indication | Interventional: 6 R-CHOP-21 for Patients Without Radiotherapy Indication | Interventional: 6 R-CHOP-14 for Patients Without Radiotherapy Indication
All-Cause Mortality (participants affected / at risk) | 7/81 | 7/81 | 15/155 | 11/150 | 10/114 | 11/114
Serious Adverse Events (participants affected / at risk) | 17/81 | 17/81 | 43/155 | 41/150 | 30/114 | 27/114
Other Adverse Events (participants affected / at risk) | 49/81 | 58/81 | 98/155 | 82/150 | 41/114 | 65/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Interventional: 6 R-CHOP-21 for Patients With Radiotherapy Indication (N=81) | Interventional: 6 R-CHOP-14 for Patients With Radiotherapy Indication (N=81) | Interventional: 6 R-CHOP-21 + Radiotherapy for Patients With Radiotherapy Indication (N=155) | Interventional: 6 R-CHOP-14 + Radiotherapy for Patients With Radiotherapy Indication (N=150) | Interventional: 6 R-CHOP-21 for Patients Without Radiotherapy Indication (N=114) | Interventional: 6 R-CHOP-14 for Patients Without Radiotherapy Indication (N=114)
Life-threatening infections (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Severe Cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
secondary neoplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1 | 7 | 4 | 8 | 8
unplanned hospitalisation (emergency case) (General disorders) | 10 (14) | 14 (17) | 28 (36) | 27 (37) | 17 (20) | 16 (25)
other (General disorders) | 1 (2) | 2 (2) | 7 (7) | 7 (7) | 5 (5) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Interventional: 6 R-CHOP-21 for Patients With Radiotherapy Indication (N=81) | Interventional: 6 R-CHOP-14 for Patients With Radiotherapy Indication (N=81) | Interventional: 6 R-CHOP-21 + Radiotherapy for Patients With Radiotherapy Indication (N=155) | Interventional: 6 R-CHOP-14 + Radiotherapy for Patients With Radiotherapy Indication (N=150) | Interventional: 6 R-CHOP-21 for Patients Without Radiotherapy Indication (N=114) | Interventional: 6 R-CHOP-14 for Patients Without Radiotherapy Indication (N=114)
Nausea CTC 3-5 (Gastrointestinal disorders) | 1/75 | 5/75 | 7/148 | 5/138 | 1/105 | 3/112 — due to limited documentation (missing data) in the database the number of paticipants at risk for each adverse event is less than the total number of participants at risk
Vomiting CTC 3-5 (Gastrointestinal disorders) | 1/74 | 3/75 | 4/148 | 2/137 | 2/105 | 1/112 — due to limited documentation (missing data) in the database the number of paticipants at risk for each adverse event is less than the total number of participants at risk
Diarrhoe CTC 3-5 (Gastrointestinal disorders) | 0/76 | 1/75 | 2/149 | 1/139 | 0/105 | 1/112 — due to limited documentation (missing data) in the database the number of paticipants at risk for each adverse event is less than the total number of participants at risk
Arrhythmia CTC 3-5 (Cardiac disorders) | 0/75 | 0/74 | 0/149 | 2/141 | 2/105 | 0/112 — due to limited documentation (missing data) in the database the number of paticipants at risk for each adverse event is less than the total number of participants at risk
Cardiac functions CTC 3-5 (Cardiac disorders) | 0/73 | 0/72 | 1/149 | 2/138 | 0/105 | 0/112 — due to limited documentation (missing data) in the database the number of paticipants at risk for each adverse event is less than the total number of participants at risk
Sensory CTC 3-5 (Nervous system disorders) | 3/75 | 4/76 | 10/150 | 4/141 | 3/103 | 8/111 — due to limited documentation (missing data) in the database the number of paticipants at risk for each adverse event is less than the total number of participants at risk
Infection CTC 3-5 (Infections and infestations) | 6/79 | 12/78 | 13/152 | 15/144 | 8/105 | 12/113 — due to limited documentation (missing data) in the database the number of paticipants at risk for each adverse event is less than the total number of participants at risk
Constipation CTC 3-5 (Gastrointestinal disorders) | 1/75 | 0/74 | 2/148 | 2/139 | 0/105 | 2/112 — due to limited documentation (missing data) in the database the number of paticipants at risk for each adverse event is less than the total number of participants at risk
Mucositis CTC 3-5 (Infections and infestations) | 0/76 | 1/75 | 0/149 | 1/140 | 0/105 | 3/112 — due to limited documentation (missing data) in the database the number of paticipants at risk for each adverse event is less than the total number of participants at risk
Mood CTC 3-5 (Psychiatric disorders) | 0/74 | 0/75 | 1/148 | 0/139 | 0/105 | 1/112 — due to limited documentation (missing data) in the database the number of paticipants at risk for each adverse event is less than the total number of participants at risk
Allergy CTC 3-5 (Immune system disorders) | 2/75 | 4/75 | 1/149 | 3/139 | 0/105 | 1/113 — due to limited documentation (missing data) in the database the number of paticipants at risk for each adverse event is less than the total number of participants at risk
Leukocytopenia CTC 3, 4 (Blood and lymphatic system disorders) | 31/43 | 22/44 | 45/76 | 36/83 | 21/49 | 21/55
Thrombocytopenia CTC 3, 4 (Blood and lymphatic system disorders) | 3/76 | 3/75 | 3/142 | 0/137 | 2/99 | 1/103
Anemia CTC 3, 4 (Blood and lymphatic system disorders) | 1/76 | 3/76 | 9/145 | 10/136 | 2/100 | 11/104

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Regarding publications the PIs and the sponsor will be in understanding between considering the publication arrangement of the trial protocol. This only serves the optimization of the research activity and the security of the results for the community.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2013-02-25): https://cdn.clinicaltrials.gov/large-docs/08/NCT00278408/Prot_SAP_ICF_000.pdf